CLINICAL TRIAL: NCT00709098
Title: A Multicenter, Double-blind, Randomized Study Comparing the Safety and Tolerability of Iloprost Inhalation Solution Delivered by I-neb Utilizing Power Disc-15 and Power Disc-6 in Patients With Symptomatic Pulmonary Arterial Hypertension
Brief Title: Safety Study Extension of Iloprost Power 15 in Pulmonary Arterial Hypertension
Acronym: PROWESS 15 Ext
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AC-063A302
Record Dates: First submitted 2008-07-01; First posted 2008-07-03 (Estimated); Results first posted 2012-10-29 (Estimated); Last update posted 2015-09-28 (Estimated); Status verified 2015-03

CONDITIONS: Pulmonary Arterial Hypertension
Keywords: pulmonary arterial hypertension; inhaled treatment; inhalation solution; iloprost; Ventavis
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — Iloprost

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- iloprost power 6 (Active Comparator): iloprost power 15
  Interventions: Drug: iloprost
- iloprost power 15 (Experimental): iloprost power 15
  Interventions: Drug: iloprost

INTERVENTIONS:
Drug: iloprost — Iloprost 5 mcg delivered by I-neb(R) adaptive aerosol delivery (AAD)(R) System power disc-6 administered 6 to 9 times per day for 12 weeks. If patient enters open label follow-up period, iloprost 5 mcg delivered by I-neb(R)AAD(R) System power disc-15 administered 6 to 9 times per day until the end of study.
  Other Names: Ventavis
  Arms: iloprost power 6
Drug: iloprost — Iloprost 5 mcg delivered by I-neb(R)AAD(R) System power disc-15 administered 6 to 9 times per day for 12 weeks. If patient enters open label follow-up period, iloprost 5 mcg delivered by I-neb(R)AAD(R) System power disc-15 administered 6 to 9 times per day until the end of study.
  Other Names: Ventavis
  Arms: iloprost power 15

SUMMARY:
Patients with symptomatic idiopathic (IPAH) or familial (FPAH) pulmonary arterial hypertension in New York Heart Association (NYHA) class II to IV , naive to PAH treatment or currently being treated with a stable dose of either bosentan or sildenafil and who complete PROWESS 15 will be enrolled in the PROWESS 15 Extension study. This is a double-blind (12 week), randomized study to compare the safety and tolerability of inhaled iloprost power disc-15 and power disc-6 in patients with symptomatic pulmonary arterial hypertension (PAH). After completion of the double blind period, patients will be entered in the open label period using iloprost power disc-15.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent prior to initiation of any study mandated procedure,
2. Patients with symptomatic idiopathic or familial pulmonary arterial hypertension in NYHA functional class II to IV who have completed study AC-063A301,
3. Women of childbearing potential must have a negative urine pregnancy test and must use an adequate method of contraception during the study and for 28 days after discontinuation of the study drug.

Exclusion Criteria:

1. Pulmonary arterial hypertension related to any condition other than those specified in the inclusion criteria,
2. Pulmonary arterial hypertension associated with significant venous or capillary involvement (Pulmonary capillary wedge pressure (PCWP) > 15 mmHg), known pulmonary veno-occlusive disease, or pulmonary capillary hemangiomatosis,
3. Moderate to severe obstructive lung disease: forced expiratory volume in 1 second/forced vital capacity (FEV1/FVC) < 70% and FEV1 < 65% of predicted value after bronchodilator administration,
4. Moderate to severe restrictive lung disease: total lung capacity (TLC) < 60% of predicted value,
5. Pregnant or breast-feeding women,
6. Systemic hypertension (systolic blood pressure > 160 mmHg or diastolic blood pressure > 100 mmHg on repeated measurement),
7. Systolic blood pressure < 95 mmHg,
8. Moderate to severe hepatic impairment, i.e., Child-Pugh Class B or C,
9. Chronic renal insufficiency defined by serum creatinine > 2.5 mg/dL (221 μmol/L) or ongoing dialysis,
10. Clinically relevant bleeding disorder or active bleeding,
11. Known hypersensitivity to iloprost or any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2008-09; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laila Rouault, MD, Study Director — Actelion
Locations (34):
- United States (32):
  - UCSD Medical Center, La Jolla, California
  - UC Davis Medical Center, Sacramento, California
  - Liu Center for Pulmonary Hypertension - LA Biomedical Research Institute at Harbor-UCLA, Torrance, California
  - Lung Health & Sleep Enhancement Center, LLC, Newark, Delaware
  - University of Florida, Gainesville, Florida
  - Pulmonary & Critical Care of Atlanta, Atlanta, Georgia
  - Atlanta Institute for Medical Research, Decatur, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Hospital, Iowa City, Iowa
  - Kentuckiana Pulmonary Associates, Louisville, Kentucky
  - LSU Health Sciences Center, New Orleans, Louisiana
  - University of Maryland Medical Center, Baltimore, Maryland
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Winthrop University Hospital, Mineola, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - The Lindner Clinical Trial Center, Cincinnati, Ohio
  - The Ohio State University Medical Center, Columbus, Ohio
  - Legacy Health System, Portland, Oregon
  - Temple University Hospital, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - Rhode Island Hospital, Providence, Rhode Island
  - Lexington Pulmonary & Critical Care, Lexington, South Carolina
  - UT Southwestern Medical Center Heart Lung and Vacular Center, Dallas, Texas
  - University of Texas Medical School, Houston, Texas
  - Central Utah Clinic, P.C., American Fork, Utah
  - Intermountain Medical Center, Murray, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Hospitals T/A Sentara Cardiovascular Research Institute, Norfolk, Virginia
  - Spokane Respiratory Consultants, Spokane, Washington
  - UW Hospital & Clinics, Madison, Wisconsin
  - Comprehensive Cardiovascular Care LLP, Milwaukee, Wisconsin
- LHK Universitatsklinikum Graz, Graz, Austria
- Universitatsklinikum Carl-Gustav-Carus, Dresden, Germany

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The double-blind period of the study was conducted at 20 centers in the US and Germany, and the following open-label period of the study was conducted at 17 centers in the US only. First patient, first visit was 4 September 2008 and the last patient, last visit was 17 June 2010.
Pre-assignment Details: Out of the 63 patients who completed the core study of AC-063A301, 49 gave informed consent and enrolled into this extension study.
Groups:
- Iloprost Power 6 (Double-blind Period): The study medication was 5 μg iloprost delivered as an aerosol using the I-neb® adaptive aerosol delivery (AAD®) System utilizing a power setting 6 disc
- Iloprost Power 15 (Double-blind Period); Iloprost Power 15 (Open-label Period): The study medication was 5 μg iloprost delivered as an aerosol using the I-neb®AAD® System utilizing a power setting 15 disc
Period: Double-blind Period
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Started | 25 | 24 | 0
Completed | 19 | 16 | 0
Not Completed | 6 | 8 | 0
Not completed — Withdrawal of consent | 3 | 3 | 0
Not completed — Administrative reason | 1 | 3 | 0
Not completed — Death | 1 | 1 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Period: Open-label Period
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Started | 0 | 0 | 32 (The open-label period was only made available to patients in US centers)
Completed | 0 | 0 | 18
Not Completed | 0 | 0 | 14
Not completed — Withdrawal of consent | 0 | 0 | 7
Not completed — Administrative reason | 0 | 0 | 5
Not completed — Death | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period) | Total
Number analyzed (Participants) | 25 | 24 | 0 | 49
Age, Continuous [Mean (Full Range); unit: years] | 58.3 (16.49) [25 to 87] | 55.4 (13.96) [29 to 79] |  | 56.9 (15.21) [25 to 87]
Gender [Number; unit: participants]
  Female | 19 | 19 |  | 38
  Male | 6 | 5 |  | 11
Region of Enrollment [Number; unit: participants]
  United States | 23 | 22 |  | 45
  Germany | 2 | 2 |  | 4

OUTCOME MEASURES:

1. Primary Outcome: Treatment-emergent Adverse Events
Description: Number of adverse events
Time Frame: Double-blind period: from first inhalation of study drug to end of 12-week treatment period. Open-label period: from the start to end of open-label medication, mean duration of exposure was 284.5 days.
Population: Safety population
Measure: Number; unit: adverse events
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Number analyzed (Participants) | 25 | 24 | 32
adverse events | 148 | 139 | 126

2. Primary Outcome: Treatment-emergent Serious Adverse Events
Description: Number of serious adverse events
Time Frame: as for outcome 1
Population: Safety population
Measure: Number; unit: serious adverse events
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Number analyzed (Participants) | 25 | 24 | 32
serious adverse events | 11 | 11 | 10

3. Primary Outcome: Adverse Events Leading to Premature Discontinuation of Study Drug
Description: Number of adverse events leading to discontinuation of study treatment
Time Frame: Double-blind period: from the first inhalation of study drug to discontinuation. Open-label period: from the start of open-label medication to discontinuation, mean duration of exposure was 284.5 days.
Population: Safety population
Measure: Number; unit: adverse events
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Number analyzed (Participants) | 25 | 24 | 32
adverse events | 3 | 10 | 7

4. Primary Outcome: Patients With Adverse Events Leading to Premature Discontinuation of Study Drug
Description: Number of patients with adverse events leading to discontinuation of study treatment
Time Frame: as for outcome 3
Measure: Number; unit: participants
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Number analyzed (Participants) | 25 | 24 | 32
participants | 2 | 6 | 7

5. Other Pre Specified Outcome: Average Inhalation Time
Description: Average inhalation time of iloprost during the double-blind period (i.e., the sum of the duration of each inhalation divided by the number of inhalations during the double-blind period)
Time Frame: 12 weeks
Population: All treated population
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Iloprost Power 6 (Double-blind Period): The study medication was 5 μg iloprost delivered as an aerosol using the I-neb®AAD® System utilizing a power setting 6 disc
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period)
Number analyzed (Participants) | 25 | 24
minutes | 10.9 (4.50) | 5.8 (1.14)
Statistical Analysis 1: Comparison: Iloprost Power 6 (Double-blind Period) vs Iloprost Power 15 (Double-blind Period); Test type: Superiority or Other; p < 0.0001, t-test, 2 sided; Mean group difference = -5.1, 95% CI 2-sided [-7.0 to -3.1]

ADVERSE EVENTS:
Time Frame: Double-blind period: from first inhalation of study drug to end of 12-week treatment period. Open-label period: from the start to end of open-label medication
Description: Treatment-emergent adverse events
Arm/Group | Iloprost Power 6 (Double-blind Period) | Iloprost Power 15 (Double-blind Period) | Iloprost Power 15 (Open-label Period)
Serious Adverse Events (participants affected / at risk) | 6/25 | 5/24 | 8/32
Other Adverse Events (participants affected / at risk) | 23/25 | 23/24 | 25/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost Power 6 (Double-blind Period) (N=25) | Iloprost Power 15 (Double-blind Period) (N=24) | Iloprost Power 15 (Open-label Period) (N=32)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 | 1 | 0
ATRIAL FLUTTER (Cardiac disorders) | 0 | 1 | 0
BRONCHITIS (Infections and infestations) | 1 | 0 | 1
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 | 0 | 0
CHOLECYSTITIS ACUTE (Hepatobiliary disorders) | 1 | 0 | 0
CHRONIC OBSTRUCTIVE PULMONARY DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
COLITIS (Gastrointestinal disorders) | 0 | 1 | 0
DIVERTICULITIS (Infections and infestations) | 1 | 0 | 0
DIVERTICULUM (Gastrointestinal disorders) | 1 | 0 | 0
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
LIVER FUNCTION TEST ABNORMAL (Investigations) | 0 | 1 | 0
LOBAR PNEUMONIA (Infections and infestations) | 1 | 0 | 0
PERIPHERAL VASCULAR DISORDER (Vascular disorders) | 0 | 1 | 0
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1
RENAL FAILURE ACUTE (Renal and urinary disorders) | 0 | 1 | 0
RESPIRATORY FAILURE (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
RIGHT VENTRICULAR FAILURE (Cardiac disorders) | 1 | 0 | 0
SEPSIS (Infections and infestations) | 0 | 1 | 0
SUDDEN CARDIAC DEATH (General disorders) | 1 | 0 | 0
SYNCOPE (Nervous system disorders) | 1 | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1 | 0
PULMONARY ARTERIAL HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 3
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
NO THERAPEUTIC RESPONSE (General disorders) | 0 | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Iloprost Power 6 (Double-blind Period) (N=25) | Iloprost Power 15 (Double-blind Period) (N=24) | Iloprost Power 15 (Open-label Period) (N=32)
HEADACHE (Nervous system disorders) | 11 | 13 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 7 | 10 | 2
DIZZINESS (Nervous system disorders) | 8 | 7 | 4
FLUSHING (Vascular disorders) | 6 | 8 | 0
NAUSEA (Gastrointestinal disorders) | 6 | 5 | 5
CHEST DISCOMFORT (General disorders) | 6 | 4 | 0
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 5 | 3 | 5
DIARRHOEA (Gastrointestinal disorders) | 3 | 4 | 5
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 3
CHEST PAIN (General disorders) | 2 | 4 | 2
FATIGUE (General disorders) | 1 | 4 | 2
PAIN IN JAW (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2 | 0
DEPRESSION (Psychiatric disorders) | 2 | 2 | 0
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 0
VOMITING (Gastrointestinal disorders) | 4 | 0 | 3
ASTHENIA (General disorders) | 2 | 1 | 0
NASOPHARYNGITIS (Infections and infestations) | 2 | 1 | 0
SYNCOPE (Nervous system disorders) | 0 | 3 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3
OEDEMA PERIPHERAL (General disorders) | 0 | 0 | 3
PALPITATIONS (Cardiac disorders) | 0 | 0 | 3
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 | 0 | 2
ACUTE SINUSITIS (Infections and infestations) | 0 | 0 | 2
ANXIETY (Psychiatric disorders) | 0 | 0 | 2
BRONCHITIS (Infections and infestations) | 0 | 0 | 2
DYSPNOEA EXERTIONAL (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
EAR INFECTION (Infections and infestations) | 0 | 0 | 2
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
INFLUENZA (Infections and infestations) | 0 | 0 | 2
INSOMNIA (Psychiatric disorders) | 0 | 0 | 2
SINUSITIS (Infections and infestations) | 0 | 0 | 2
URINARY TRACT INFECTION (Infections and infestations) | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No